CLINICAL TRIAL: NCT03081533
Title: Brazilian Circle Dance Program for Family Caregivers of the Elderly With Alzheimer's Disease (CircleCare): a Single-blind, Parallel-group Randomized Controlled Trial
Brief Title: Circle Dance for Family Caregivers of the Elderly With Alzheimer.
Acronym: CircleCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Julimara Gomes dos Santos, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 62112716.8.0000.5504
Record Dates: First submitted 2017-03-02; First posted 2017-03-16 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Family Caregiver
Keywords: Healthy Aging; Family Health; Exercise; Dance Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will be blind to groups allocation (experimental and control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circle Dance Program (CircleCare) (Experimental): Caregivers (n=20) allocated to the experimental group will participate in 12-week CircleCare twice a week (24 sessions), for 60 min each session. The planning and conduction of the intervention will be the responsibility of the researcher, a Fitness Professional with training in Circle Dance, called focalizer.
  Interventions: Other: Circle Dance Program (CircleCare)
- Control group (No Intervention): Caregivers (n=20) of this group will not receive the intervention, participating only in the assessment protocol. They will be instructed not to initiate any regular exercise program during the study period. At the end of the study, the same CircleCare applied to the experimental group will be offered to the interested of the control group.

INTERVENTIONS:
Other: Circle Dance Program (CircleCare) — Circle Dances derives from folk dances, but their current repertoire encompasses traditional and contemporary dances from diverse nations and cultures around the world. Most of the choreographies are danced with the participants placed in a circle, holding hands, repeating a pattern of steps to the rhythm of the music.
  Other Names: Dance
  Arms: Circle Dance Program (CircleCare)

SUMMARY:
The primary objective of this research is to compare the effects of a 12-week CircleCare on physical functioning of family caregivers of the elderly with AD. Effects on cognition, psychosocial and frailty-related aspects (secondary objective). The acute effect of one circle dance session on mood states (tertiary objective). This randomized controlled trial will involve 40 family caregivers over 50 years old allocated into a control group or an intervention group of 12-weeks (twice a week, 60 min per session) of CircleCare. Primary outcomes will include balance, speed of gait, lower limb muscle strength, functional mobility and risk of falls. Secondary outcomes will include cognition, burden, stress, depression, quality of life and frailty. Mood states will be a tertiary outcome. The effects of CircleCare will be verified with an ANOVA two-way test and a multiple comparison test when necessary. The analyzes will follow an intention-to-treat approach. The change in moods will be evaluated by the paired t-test. The level of significance will be set at p<0.05. This study may guide professionals and health policymakers in deciding whether to implement this type of intervention. If positive effects are demonstrated, this program can be offered in public health services to other groups, given its low cost.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older.
* Family caregiver for at least 6 months of an elderly person with Alzheimer's disease.
* Ability to walk without the help of another person.

Exclusion Criteria:

* Cardiopulmonary or orthopaedic contraindication to the practice of physical exercise.
* Severe visual or hearing deficiency that impedes participation in the intervention and assessments.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-06-14 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Brazilian Version of the Short Physical Performance Battery | Baseline and 12 weeks after randomization.
  Battery tests that evaluate the static balance; the speed of gait and lower limb muscle strength. Each test ranges from zero to four points, and the total score is obtained by summing the score of each test, ranging from zero to 12 points. The result can receive the following graduation: 0 to 3 points: incapacity or very poor performance; 4 to 6 points: low performance; 7 to 9 points: moderate performance; 10 to 12 points: good performance.
Timed Up and Go Test | Baseline and 12 weeks after randomization.
  Test that evaluates the basic functional mobility through the time spent to get up from a chair with arms, walk 3 meters and return to the chair, as well as the number of steps required to perform the activity. The shorter the time to perform the task, the better the mobility index. The 12.47 second cutoff point will be used as an indicator of the risk of falls.

SECONDARY OUTCOMES:
Addenbrooke's Cognitive Examination-Revised (ACE-R) | Baseline and 12 weeks after randomization
  Portuguese version of the Instrument that evaluates the global cognitive function through individual tests of orientation and attention (18 points), memory (26 points), verbal fluency (14 points), language (26 points) and spatial visibility skills (16 points). The overall score ranges from zero to 100 points.
Zarit Burden Interview (ZBI) | Baseline and 12 weeks after randomization
  An instrument that evaluates the physical, psychological and social impact of the task of caring for a patient with mental illness. The scale is composed of 22 questions, whose scores can range from 0 to 88 points. A score below 21 points is classified as no burden; of 21 and 40 points indicate a moderate burden; between 41 to 60, moderate to severe burden and ≥ 61 points, a severe burden.
Brazilian Perceived Stress Scale (BPSS-10) | Baseline and 12 weeks after randomization
  PSS-10 is used to assess the level of stress perceived by older adults in the last month. The final score ranges from 0 to 40, with higher scores denoting a greater degree of perceived stress.
Geriatric Depression Scale (GDS-15) | Baseline and 12 weeks after randomization
  Scale composed of 15 negative/affirmative questions that evaluate the presence of depressive symptoms in the elderly. Scores higher than 5 points indicate the risk of depression.
Quality of Life Scale in Alzheimer's disease (QoL-AD - caregiver's version) | Baseline and 12 weeks after randomization
  Scale structured in three versions that relate to the quality of life of the elderly, careAn instrument adapted, translated and validated for the Brazilian culture to assess the quality of life of caregivers and elderly with AD. In this version the caregiver to assess his/her own quality of life. The score ranges from 13 to 52 points and the lower the score worse is the quality of life.
Frailty Phenotype | Baseline and 12 weeks after randomization
  A battery of tests proposed by Fried et al. (2001) that asses unintentional weight loss (10 lbs in the past year), self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity. Participants with three or more criteria will be classified as frail. Those with one or two criteria, pre-frail. "No frail" will correspond to the absence of these criteria.

OTHER OUTCOMES:
Illustrated and Reduced Mood States List (MSL-IR) | After randomization, at the beginning and end of the first CircleCare session.
  Scale that evaluates the intensity of positive and negative moods represented by 14 "smile" faces.

CONTACTS AND LOCATIONS:
Locations (1):
- Julimara Gomes dos Santos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
At the end of the study, caregivers will be individually informed about their performance in the assessments, but your personal data will not be shared with others, respecting your privacy and anonymity. However, the analyzed results will be published in papers, reported in congresses and special interest groups such as groups of Alzheimer's caregivers and health units interested in implementing the circle dances as a health promotion activity.